CLINICAL TRIAL: NCT06773715
Title: Changing the View of Pain: Using Virtual Reality As Adjunctive Therapy for Sickle Cell Pain in Pediatric Patients
Brief Title: Virtual Reality As Adjunct Therapy for Vaso-Occlusive Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: KindVR (Unknown)
Responsible Party: Principal Investigator, Molly Sonenklar, Assistant Professor in Pediatrics, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB# 7634
Record Dates: First submitted 2024-11-14; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Pain Episodes
Keywords: virtual reality; adjunctive therapy; opiate consumption; pain reduction
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
  * Control patients will receive standard of care therapy for their vaso-occlusive pain crisis
  * Case patients will receive standard of care therapy PLUS VR experience for their vaso-occlusive pain crisis
  * Patients will be randomly assigned into the case or control group based off a random number system that will assign N/2 patients into each group. The statistician included on this project will generate the random numbers prior to the enrollment of the first patient onto the study.
  * To ensure equality between case and control groups, block stratification based on age and gender will be utilized at the time of data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controls (No Intervention): Control patients will continue to receive the standard of care for their vaso-occlusive pain (IV fluid hydration, scheduled IV NSAID, and opiate medication) and have repeat pain assessments at 1 hour and 4 hours from their baseline assessment. This same timeline will occur on days 2 and 3 of admission
- Cases (Experimental): In addition to receiving the standard of care for their vaso-occlusive pain, the case patients will have the opportunity to participate in the immersive VR experience after completing their initial pain assessment simulator sickness survey. Following the intervention, their pain levels will be reassessed at the 1-hour and 4-hour mark from their baseline assessment. Additionally, they will be asked to fill out an additional simulator sickness survey upon completion of the VR experience. This same timeline will occur on days 2 and 3 of admission. Prior to discharge or discontinuation from the study, the case patients will be asked to fill out the post-study questionnaire.
  Interventions: Device: KindVR Aqua Program

INTERVENTIONS:
Device: KindVR Aqua Program — For this study, patients will be introduced to a virtual reality software program called Aqua, created by the company KindVR. This software program was designed specifically for use in pediatric patients. The software has been programmed into the Pico Neo 3 headset and provides an immersive 3D experience during which the patients explore a virtual underwater world inside a submarine with a goal of providing more color to treasure and different sea animals that they will engage with along their journey. The VR experience itself lasts approximately 15 minutes
  Arms: Cases

SUMMARY:
The goal of this randomized control clinical trial is to learn if virtual reality can be used to treat sickle cell pain in children. The main questions it aims to answer are:

Does virtual reality reduce pain severity during a child's hospital stay for a vaso-occlusive pain crisis?

Does virtual reality decrease the daily use of opiates?

Researchers will compare standard therapy to the use of standard therapy plus a daily virtual reality experience to see if virtual reality works to treat sickle cell pain.

All patients will:

- Be asked to fill out a pain assessment survey three times daily for up to 3 days

If randomized to intervention arm, patients will:

* Participate in an immersive virtual reality experience once daily for up to 3 days
* Fill out a survey twice daily to monitor for side effects from virtual reality experience
* Fill out a satisfaction survey once during the study period

DETAILED DESCRIPTION:
A vaso-occlusive pain crisis is the most common complaint for which a patient with sickle cell disease requires admission to the hospital. These pain episodes can often be complex and difficult to manage as medical providers know each individual patient perceives pain differently. In this regard, it has been well studied that a multi-disciplinary approach is required to address the biological, psychological, and social factors that comprise a patient's experienced pain. The current standard therapy for vaso-occlusive pain is heavily reliant on opioid therapy, which is why efforts have been made to find other complementary therapies with intentions of reducing this need. By conducting this study, the investigators hope to show that virtual reality can not only provide a complementary role in addressing sickle cell pain but also enhance patient satisfaction for those who have been admitted to the inpatient unit in a time of need.

The idea of using virtual reality as a complementary therapy to address pain and stress in different types of medical patients has been introduced and explored for the last 10 years. There are a limited number of studies currently being carried out, but since 2014, the KindVR company has partnered with medical institutions across the United States and Canada to study the impacts that virtual reality can have on different pediatric patients. This includes sickle cell patients experiencing a pain crisis, cancer patients undergoing port access, burn patients, and those dealing with stress associated with a procedure or imaging study. A previous study in 2018 displayed the feasibility of administering a virtual reality (VR) experience to patients admitted to the hospital for a sickle cell pain crisis. However, there are no published studies assessing the measurable impacts that the use of VR could have on aspects of patient care. It is well known that a multi-disciplinary approach is the best method to address sickle cell pain. The investigators believe it would be interesting to see if the advanced technology of virtual reality can provide a complementary role to the current standard of care.

To best elicit the results of our treatment intervention, this study will be constructed as a randomized control study. During the screening phase, every patient that is admitted to Children's Hospital of New Orleans for a vaso-occlusive pain episode will first have eligibility for enrollment into the study determined by established inclusion and exclusion criteria. Prior to enrollment, informed consent, patient assent (if applicable), and Health Insurance Portability and Accountability Act (HIPAA) authorization will be obtained. For the study treatment phase, patients will be assigned to either the control or case group. Control patients will undergo scheduled pain assessments while receiving standard of care therapy for a vaso-occlusive pain crisis. Case patients will undergo scheduled pain assessments while receiving standard of care therapy in addition to participating in a daily immersive VR experience during admission for a vaso-occlusive pain crisis. Both groups of patients will concurrently be in the hospital at the same time. All patients will participate in the study for a maximum of 3 days while enrolled on study and remain admitted requiring further treatment for vaso-occlusive pain. There will be no follow-up phase as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 8 up to 21 years of age
2. Presenting to CHNOLA ER or outside facility with chief complaint of vaso-occlusive pain crisis, requiring inpatient admission for further pain management
3. No known cognitive or neurological deficits
4. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Patients aged 7-years-old and younger.
2. Patents upon admission found to have sequela of their sickle cell disease that would require medical therapy greater than the standard of care for a vaso-occlusive pain event. This includes acute chest syndrome, splenic sequestration, post-operative pain, and/or cerebrovascular accident
3. Patients who are developmentally or cognitively incapable of using VR equipment and answering questions appropriately
4. Failure to obtain or refusal to provide parental/guardian permission (informed consent) and if appropriate child assent
5. Patient has previously participated in the study
6. Study team is unable to initiate study interventions within the first 24 hours of a patient's admission

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Pain severity | From enrollment to the end of hospital admission day 3.
  The Adolescent-Pediatric Pain Tool is a well validated, multidimensional pain assessment tool designed to evaluate the location, severity, and quality of pain in pediatric patients. It is comprised of three independent parts, one which is a 10 cm line anchored from 0 to10, with zero being equivalent to "no pain" and 10 being equivalent to "worst pain possible". This data point will be collected up to 9 times for each participant in this study. The trends will be compared amongst the control and case groups.

SECONDARY OUTCOMES:
Opiate Consumption | From enrollment to the end of hospital admission day 3.
  Goal is to assess virtual reality's ability to decrease a patient's total opiate consumption during their inpatient admission. Equivalent opiate dosing per day, measured in oral morphine equivalents/kg/day for each participant.
Hospital Length of Stay. | From enrollment to hospital discharge (an average of 5 days)
  Assessing whether the use of virtual reality for a patient's vaso-occlusive pain crisis can reduce their length of stay in the hospital. Measured in number of days.
Patient Satisfaction (for case patients only) | Once, on day 2 or day 3 of enrollment
  The study will evaluate whether the use of virtual reality's ability to improve patient satisfaction for their hospital admission. This will be measured via the use of the Post-Study Questionnaire, a 16-question survey provided by the KindVR company. It will be used to assess the patient's satisfaction of the Aqua program, the comfort of the equipment, and future guidance to aid quality improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litwin SP, Nguyen C, Hundert A, Stuart S, Liu D, Maguire B, Matava C, Stinson J. Virtual Reality to Reduce Procedural Pain During IV Insertion in the Pediatric Emergency Department: A Pilot Randomized Controlled Trial. Clin J Pain. 2021 Feb 1;37(2):94-101. doi: 10.1097/AJP.0000000000000894. PMID 33177370
- [Background] Fernandes AM, De Campos C, Batalha L, Perdigao A, Jacob E. Pain assessment using the adolescent pediatric pain tool: a systematic review. Pain Res Manag. 2014 Jul-Aug;19(4):212-8. doi: 10.1155/2014/979416. Epub 2014 Jun 20. PMID 24950413
- [Background] Birnie KA, Kulandaivelu Y, Jibb L, Hroch P, Positano K, Robertson S, Campbell F, Abla O, Stinson J. Usability Testing of an Interactive Virtual Reality Distraction Intervention to Reduce Procedural Pain in Children and Adolescents With Cancer [Formula: see text]. J Pediatr Oncol Nurs. 2018 Nov/Dec;35(6):406-416. doi: 10.1177/1043454218782138. Epub 2018 Jun 27. PMID 29950139
- [Background] Das DA, Grimmer KA, Sparnon AL, McRae SE, Thomas BH. The efficacy of playing a virtual reality game in modulating pain for children with acute burn injuries: a randomized controlled trial [ISRCTN87413556]. BMC Pediatr. 2005 Mar 3;5(1):1. doi: 10.1186/1471-2431-5-1. PMID 15745448
- [Background] Agrawal AK, Robertson S, Litwin L, Tringale E, Treadwell M, Hoppe C, Marsh A. Virtual reality as complementary pain therapy in hospitalized patients with sickle cell disease. Pediatr Blood Cancer. 2019 Feb;66(2):e27525. doi: 10.1002/pbc.27525. Epub 2018 Oct 26. PMID 30362236